CLINICAL TRIAL: NCT00001642
Title: Positional Cloning of the Gene(s) Responsible for Alagille Syndrome
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970122; 97-HG-0122
Record Dates: First submitted 2000-04-06; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Alagille Syndrome
Keywords: Chromosomal Deletion; Mutations; Paucity of Bile Ducts; Physical Map; Transcript Identification; Alagille Syndrome; Syndromic Bile Duct Paucity
MeSH Terms: conditions — Alagille Syndrome; Chromosome Deletion

SUMMARY:
The goal of the project is to identify and clone the gene(s) responsible for the Alagille Syndrome (AGS) by a positional cloning approach. The first step towards this goal is to define the smallest genomic candidate region for AGS at 20p12 and to begin to identify genes within this region which are, by definition, candidate genes for the disease. In a collaborative effort with clinician-investigators studying the Alagille syndrome, metaphase chromosomes and genomic DNA from affected individuals will be studied for subchromosomal deletions and for mutations in the candidate genes. Characterization of genes involved in Alagille syndrome could provide important insight into the pathophysiology of the disease, the development of normal liver and treatment of this disease. Recently, we and others found that mutations in Jagged1, a Notch1 receptor are responsible for Alagille Syndrome.

DETAILED DESCRIPTION:
The goal of the project is to identify and clone the gene(s) responsible for the Alagille Syndrome (AGS) by a positional cloning approach. The first step towards this goal is to define the smallest genomic candidate region for AGS at 20p12 and to begin to identify genes within this region which are, by definition, candidate genes for the disease. In a collaborative effort with clinician-investigators studying the Alagille syndrome, metaphase chromosomes and genomic DNA from affected individuals will be studied for subchromosomal deletions and for mutations in the candidate genes. Characterization of genes involved in Alagille syndrome could provide important insight into the pathophysiology of the disease, the development of normal liver and treatment of this disease.

ELIGIBILITY:
All enrolled affected subjects, whose samples will be analyzed in this study, must meet the criteria for the clinical diagnosis of Alagille Syndrome (Syndromic Bile Duct Paucity) which include liver biopsy findings consistent with Alagille Syndrome and at least 3 of the 5 primary clinical criteria: cholestasis, characteristic face, posterior embryotoxon, "butterfly" vertebrae and cardiac findings.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225
Dates: Start 1997-05; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Alagille D, Odievre M, Gautier M, Dommergues JP. Hepatic ductular hypoplasia associated with characteristic facies, vertebral malformations, retarded physical, mental, and sexual development, and cardiac murmur. J Pediatr. 1975 Jan;86(1):63-71. doi: 10.1016/s0022-3476(75)80706-2. PMID 803282
- [Background] Alagille D, Estrada A, Hadchouel M, Gautier M, Odievre M, Dommergues JP. Syndromic paucity of interlobular bile ducts (Alagille syndrome or arteriohepatic dysplasia): review of 80 cases. J Pediatr. 1987 Feb;110(2):195-200. doi: 10.1016/s0022-3476(87)80153-1. PMID 3806290
- [Background] Oda T, Elkahloun AG, Pike BL, Okajima K, Krantz ID, Genin A, Piccoli DA, Meltzer PS, Spinner NB, Collins FS, Chandrasekharappa SC. Mutations in the human Jagged1 gene are responsible for Alagille syndrome. Nat Genet. 1997 Jul;16(3):235-42. doi: 10.1038/ng0797-235. PMID 9207787